CLINICAL TRIAL: NCT03179527
Title: Research on the Clinical Effect of Shuanghe Decoction in Treating Unstable Angina.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jun Li (Other)
Collaborators: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Sponsor-Investigator, Jun Li, Chief Physician, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Organization: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHS-2017
Record Dates: First submitted 2017-06-05; First posted 2017-06-07 (Actual); Last update posted 2017-06-07 (Actual); Status verified 2017-06

CONDITIONS: Unstable Angina
Keywords: Unstable Angina; Shuanghe Decoction
MeSH Terms: conditions — Angina, Unstable | interventions — Lipid Regulating Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Qi deficiency and blood stasis (Experimental): Patients in this group will be treated by Shuanghe Decoction at the base of conventional western medicine.
  Interventions: Drug: Anti-Platelet Drugs; Drug: Lipid Regulating Drugs; Drug: Coronary Vasodilator; Drug: Shuanghe Decoction
- Conventional western medicine (Other): Patients in this group will be treated by conventional western medicine, including anti-platelet drugss，lipid regulating drugs, coronary vasodilator, etc.
  Interventions: Drug: Anti-Platelet Drugs; Drug: Lipid Regulating Drugs; Drug: Coronary Vasodilator

INTERVENTIONS:
Drug: Anti-Platelet Drugs — Including aspirin and clopidogrel, etc
Drug: Lipid Regulating Drugs — Mainly including statins
Drug: Coronary Vasodilator — Mainly including nitrates
Drug: Shuanghe Decoction — Mainly including Ginseng, Poria, Calamus, Cyperus, Salvia miltiorrhiza, Radix Polygalae etc.
  Arms: Qi deficiency and blood stasis

SUMMARY:
This study evaluates the clinical efficacy of Shuanghe Decoction in the treatment of unstable angina. All of the patients will be divided into 2 arms randomly. One of the arms will be treated by conventional western medicine, and the other one will be treated by Shuanghe Decoction at the base of conventional western medicine.

DETAILED DESCRIPTION:
Shuanghe Decoction has the function of supplementing Qi and activating blood circulation, which will be used to treat patients with Qi deficiency and blood stasis syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Participants diagnosed with coronary heart disease through coronary angiography or coronary CTA;

Patients have at least one of these symptoms:

1. The stability of the nature of angina pectoris changes, that is, frequent attacks of angina pectoris, serious degree and prolonged duration;
2. Angina pectoris during rest;
3. The recent occurrence of angina pectoris caused by mild physical activity in the last month.

Exclusion Criteria:

* Patients diagnosed with stable angina; Patients with acute myocardial infarction; Chest pain caused by congenital heart disease, valvular heart disease, severe neurosis or arrhythmia; The heart function grade is III or IV; Patients with acute cerebral infarction; Patients complicated with other serious primary diseases; Patients with acute infection in recent 2 weeks; Uncontrolled hypertension (the resting blood pressure >160/95mmHg within one week); Diabetics emerged with serious diabetic complications; Patients can't finish the questionnaire due to abnormal mental and nervous or mental disorders; Pregnant or lactating women.

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2017-07 (Estimated); Primary Completion 2019-10 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Mortality | Six months after drug intervention
  Death caused by cardiovascular disease

SECONDARY OUTCOMES:
Myocardial enzymes | At baseline and 4 weeks after drug intervention
  The unit is mmol/L
Blood lipid | At baseline and 4 weeks after drug intervention
  The unit is mmol/L
Treadmill exercise test | At baseline and 4 weeks after drug intervention
  The result will be positive or negative
The incidence of myocardial infarction or heart failure | Six months after drug intervention

CONTACTS AND LOCATIONS:
Overall Officials: Jun Li, MD, Study Director — Guang'anmen Hospital of China Academy of Chinese Medical Sciences

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Wang J, Yu G. A Systems Biology Approach to Characterize Biomarkers for Blood Stasis Syndrome of Unstable Angina Patients by Integrating MicroRNA and Messenger RNA Expression Profiling. Evid Based Complement Alternat Med. 2013;2013:510208. doi: 10.1155/2013/510208. Epub 2013 May 14. PMID 23762142
- [Result] Yi GZ, Qiu YQ, Xiao Y, Yuan LX. The usefulness of xuefu zhuyu tang for patients with angina pectoris: a meta-analysis and systematic review. Evid Based Complement Alternat Med. 2014;2014:521602. doi: 10.1155/2014/521602. Epub 2014 Aug 31. PMID 25254054
- [Result] Qiu Y, Xu H, Shi D. Traditional chinese herbal products for coronary heart disease: an overview of cochrane reviews. Evid Based Complement Alternat Med. 2012;2012:417387. doi: 10.1155/2012/417387. Epub 2012 Mar 28. PMID 22536282
- [Result] Liu W, Xiong X, Yang X, Chu F, Liu H. The Effect of Chinese Herbal Medicine Gualouxiebaibanxia Decoction for the Treatment of Angina Pectoris: A Systematic Review. Evid Based Complement Alternat Med. 2016;2016:8565907. doi: 10.1155/2016/8565907. Epub 2016 Sep 29. PMID 27777598
- [Result] Wang J, Yang X, Chu F, Chen J, He Q, Yao K, Teng F, Gao Y, Xing Y, Wu A, Xing Y. The effects of xuefu zhuyu and shengmai on the evolution of syndromes and inflammatory markers in patients with unstable angina pectoris after percutaneous coronary intervention: a randomised controlled clinical trial. Evid Based Complement Alternat Med. 2013;2013:896467. doi: 10.1155/2013/896467. Epub 2013 May 8. PMID 23737852